CLINICAL TRIAL: NCT05183217
Title: Tailoring Online Continence Promotion for Women
Brief Title: Tailoring Online Continence Promotion
Acronym: TOCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1555; 1R01DK128349-01 (NIH); A532800 (Other: UW Madison); Protocol Version 12/10/2021 (Other: UW Madison)
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Urinary Incontinence in Old Age; Fecal Incontinence in Old Age

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online continence promotion program without tailoring (Active Comparator): Participants will be allocated to the online continence promotion program without tailoring.
  Interventions: Behavioral: Online Continence promotion program without tailoring
- Online continence promotion program with tailoring (Experimental): Participants will be allocated to the online continence promotion program with tailoring.
  Interventions: Behavioral: Online Continence promotion program with tailoring

INTERVENTIONS:
Behavioral: Online Continence promotion program without tailoring — The online continence promotion program has five sections (Introduction, Exercise, Bladder, Bowels, Care Seeking) that build knowledge, self-efficacy, and skills to set action and coping plans relevant to a participant's symptoms. This online program is based on an in-person, small-group program that has demonstrated effectiveness to improve both urinary and bowel incontinence in women age 50 and above. Participants will receive automated weekly reminders reminding them to re-visit the program, regardless of their individual user activity.
  Other Names: Mind Over Matter; Healthy Bowels, Healthy Bladder (MOM) online without tailoring
  Arms: Online continence promotion program without tailoring
Behavioral: Online Continence promotion program with tailoring — The online continence promotion program has five sections (Introduction, Exercise, Bladder, Bowels, Care Seeking) that build knowledge, self-efficacy, and skills to set action and coping plans relevant to a participant's symptoms. This online program is based on an in-person, small-group program that has demonstrated effectiveness to improve both urinary and bowel incontinence in women age 50 and above. Participants will receive tailored "output" (personalized cues, emphasis on relevant content, individualized and tailored reminders about their goals) based on a computer algorithm incorporating unique user "inputs" (individual factors). Inputs will be reassessed every 2 weeks for retailoring so that personalization evolves over the course of the intervention.
  Other Names: Mind Over Matter; Healthy Bowels, Healthy Bladder (MOM) online with tailoring
  Arms: Online continence promotion program with tailoring

SUMMARY:
This project seeks to understand whether, and how, tailoring an online continence intervention can increase engagement and uptake of health behaviors known to improve bladder and bowel symptoms.

DETAILED DESCRIPTION:
The investigators will conduct a two-arm, parallel, randomized, controlled trial (RCT) comparing an online continence promotion program with standard weekly reminders (control arm) to an online continence promotion program with tailoring (treatment arm) to determine the impact of tailoring on program engagement. Women in the treatment arm will receive tailored content and digital reminders for 24 weeks based on their individual characteristics, symptoms, and behaviors assessed at baseline, with reassessment of key inputs every 2 weeks resulting in re-tailored outputs. Participants will complete electronic surveys at enrollment, 4, 12, and 24 weeks. To contextualize the findings from all 3 aims, a subset of participants will be invited to complete semi-structured qualitative interviews about their engagement with the program, their adoption of health behaviors, and their perceived barriers to and facilitators of engagement and behavior change.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 50 years or older
* Can read & write English
* Can use email
* Has access to an Internet-connected device to use the online program

Exclusion Criteria:

* Dementia
* Neurologic or musculoskeletal conditions in which pelvic floor muscle exercises are contraindicated
* Hematuria or bloody stools within last 6 months that has not been evaluated by a medical professional

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 445 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Piper, PhD, Principal Investigator — University of Wisconsin Dept of Medicine
Locations (1):
- University of Wisconsin-Madison School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Online Continence Promotion Program Without Tailoring | Online Continence Promotion Program With Tailoring
Started | 226 | 219
Completed | 225 | 218
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Online Continence Promotion Program Without Tailoring | Online Continence Promotion Program With Tailoring | Total
Number analyzed (Participants) | 226 | 219 | 445
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 58 [54 to 65] | 58 [54 to 63] | 58 [54 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226 | 219 | 445
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 219 | 212 | 431
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 6
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 41 | 34 | 75
  White | 174 | 175 | 349
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 226 | 219 | 444
Height [Median (Inter-Quartile Range); unit: Centimeters] | 165 [160 to 170] | 165 [160 to 170] | 165 [160 to 170]
Weight [Median (Inter-Quartile Range); unit: kilograms] | 77 [64 to 93] | 75 [63 to 89] | 76 [63 to 93]
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 28 [24 to 33] | 27 [23 to 32] | 27.5 [23 to 33]

OUTCOME MEASURES:

1. Primary Outcome: User Engagement With Online Mind Over Matter (MOM)
Description: Proportion of participants who engage with online MOM at least 4 times during weeks 0-4 in the group with (test) and without (control) tailoring.
Time Frame: 0-4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Online Continence Promotion Program Without Tailoring | Online Continence Promotion Program With Tailoring
Number analyzed (Participants) | 226 | 219
Participants | 17 | 37

2. Secondary Outcome: Self-reported Behavior Changes: Change in the Frequency of Pelvic Floor Muscle Exercises
Description: Frequency of pelvic floor muscle exercises
Time Frame: Baseline, 4, 12, and 24 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Differences in Scores of the Geriatric Index for Urinary Incontinence (GSE-UI)
Description: The Geriatric Index for Urinary Incontinence (GSE-UI) is a validated and clinically responsive instrument for older women with urinary incontinence. Participants select a 0-10 score for each of the 12 items, with total scores ranging from 0-120. A higher score is indicative of a higher level of self-efficacy related to urinary incontinence.
Time Frame: Baseline, 4, and 24 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Differences in Responses to the Generalized Self-Efficacy Scale Adapted for MOM Program
Description: Previously, in consultation with Dr. Ralf Schwarzer (Health Action Process Approach developer), the investigators adapted the Generalized Self Efficacy scale for behaviors related to continence promotion (such as pelvic floor muscle exercises).10-items are scored on a 4 point likert scale from 1 (not true at all) to 4 (exactly true) for a total range of scores from 10-40 where higher scores indicate higher self-efficacy.
Time Frame: Baseline, 4, and 24 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Program Specific Health Action Process Approach Survey Responses Reported as Binary Outcomes
Description: Number of Participants who report high vs low risk perception, positive vs negative outcome expectations, specific intentions, action or coping plans, barriers and facilitators for health on the program-specific survey of other Health Action Process Approach components.
Time Frame: Baseline, 4, and 24 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Differences in Scores of the Barriers to Incontinence Care-Seeking Questionnaire (BICS-Q)
Description: The Barriers to Incontinence Care-Seeking Questionnaire (BICS-Q) contains 14-items framed on a 4-point Likert scale and is validated in women with urinary incontinence. Mean score will be reported, ranging from 1-4 where higher scores indicate increased barriers.
Time Frame: Baseline and 24 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Differences in Scores of the Barriers to Care-seeking for Accidental Bowel Leakage (BCABL)
Description: The Barriers to Care-seeking for Accidental Bowel Leakage (BCABL) has been validated in women with bowel incontinence. BCABL contains 16 questions framed on a 4-point Likert scale (strongly disagree, somewhat disagree, somewhat agree, strongly agree), for a total possible range of scores from 16-64 where higher scores indicate increased barriers.
Time Frame: Baseline and 24 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Differences in Scores of the International Consultation on Incontinence Questionnaire-Urinary Incontinence (ICIQ-UI)
Description: ICIQ-UI is a subjective measure of severity of urinary loss and quality of life for those with urinary incontinence. It is scored on a scale from 0-21. Based on the score participant can be placed in four severity categories: slight (1-5), moderate (6-12), severe (13-18) and very severe (19-21)
Time Frame: Baseline, 4, 12, and 24 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Differences in Scores of the St. Mark's Incontinence Scale (SMIS) (Aka Vaizey)
Description: St. Mark's Incontinence Scale (aka Vaizey) will be used to assess the severity and the outcome of MOM intervention
  Never: no episodes in the past 4 weeks rarely: 1 episode in the past 4 weeks sometimes: > 1 episode in the past 4 weeks, but,1 a week; Weekly: 1 or more episodes a week but,1 a day Daily: 1 or more episodes a day
  Scores will be assigned for each row (Never=0, Rarely=1, Sometimes=2, Weekly=3, Daily=4 )
  Score will be added from each row. Cumulative minimum score=0 perfect continence; Cumulative maximum score will be 24= totally incontinence
Time Frame: Baseline, 4, 12, and 24 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Differences in Scores of the Pelvic Floor Impact Questionnaire Short Form (PFIQ-7)
Description: The Pelvic Floor Impact Questionnaire Short Form (PFIQ-7) is a widely-used validated instrument that assesses condition-specific quality of life. Scores range from 0-300 with higher scores indicating higher symptom bother.
Time Frame: Baseline, 4, 12, and 24 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Change in the Response of Global Patient Satisfaction Question (PSQ)
Description: Patient satisfaction will be measured with the question: How satisfied are you with your progress in this program? (completely, some-what, not at all)
Time Frame: 4 and 24 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Change in Patient Estimated Percent Improvement (EPI)
Description: For EPI, Patients will be asked to estimate how much better they were on a scale from 0% (no better) to 100%(completely better)
Time Frame: 4 and 24 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Change in Response on Global Perception of Improvement (GPI)
Description: Global perception of improvement (GPI) is a tool for Global Rating of Patient Satisfaction and Perceptions of Improvement.
  Question asked: Overall, do you feel that you are? Response can be chosen from the options: Much Better, Better, About the same, Worse, Much worse
Time Frame: 4 and 24 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Differences in Scores of the 12-item Short Form Health Survey (SF-12)
Description: The 12-item Short Form Health Survey (SF-12) is a validated health-related quality of life questionnaire from which mental and physical component scores can be calculated. Scores on the PCS-12 (Physical Score): range from 23.99938 (difference from USA average: -26.00062) to 56.57706 (difference from USA average: 6.57706). Scores on the MCS-12 (Mental Score): range from 19.06444 (difference from USA average: -30.93556) to 60.75781 (difference from USA average: 10.75781). For both components, higher scores indicate better health-related quality of life.
Time Frame: Baseline, 4, 12, and 24 weeks
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Program Use Metrics
Description: Comparison of specific program use metrics (number of, minutes spent on, and average intervals between program sessions accessed weekly; number of and specific components accessed) between the two groups and patterns of program use (such as tracking and reminders).
Time Frame: Baseline to 24 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Self-reported Behavior Changes: Change in Body Mass Index (BMI)
Description: Proportion of participants in the treatment group compared to the control group with a body mass index (BMI) >25mg/kg2 at baseline who report weight loss of at least 2 kg.
Time Frame: Baseline, 4, 12, and 24 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Self-reported Behavior Changes: Change in Fluid Intake
Description: Self-reported behavior changes: fluid intake
Time Frame: Baseline, 4, 12, and 24 weeks
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Self-reported Behavior Changes: Change in Fiber Intake
Description: Self-reported behavior changes: change in fiber intake
Time Frame: Baseline, 4, 12, and 24 weeks
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Self-reported Coping Changes: Change in Types of Pad Used
Description: Self-reported coping changes: change in types of pad used
Time Frame: Baseline, 4, 12, and 24 weeks
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Self-reported Coping Changes: Change in Number of Pads Used
Description: Self-reported coping changes: change in number of pads used
Time Frame: Baseline, 4, 12, and 24 weeks
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Self-reported Changes: Change in the Money-spent on Buying Products to Manage Their Incontinence
Description: It will be measured by asking participants question that how much money have they spent on products (such as pads, undergarments, or plugs) to manage their bladder and/or bowel symptoms in the last month.
Time Frame: Baseline, 4, 12, and 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Online Continence Promotion Program Without Tailoring | Online Continence Promotion Program With Tailoring
All-Cause Mortality (participants affected / at risk) | 0/225 | 0/219
Serious Adverse Events (participants affected / at risk) | 0/225 | 0/219
Other Adverse Events (participants affected / at risk) | 0/225 | 0/219

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT05183217/Prot_SAP_001.pdf
  • Informed Consent Form (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT05183217/ICF_000.pdf